CLINICAL TRIAL: NCT03084198
Title: Safety and Efficacy of hiHep Bioartificial Liver Support System to Treat Acute Liver Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai East Hospital (Other)
Collaborators: Chinese Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFSC-2015（CR）-05
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Liver Failure, Acute
Keywords: Bioartificial Liver; Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute | interventions — Standard of Care; GTF2A1L protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Standard care for ALF
  Interventions: Procedure: Standard care for ALF
- Experimental group (Experimental): Continuous treatment with the hiHep bioartificial liver support system.
  Interventions: Procedure: hiHep Bioartificial Liver Support System

INTERVENTIONS:
Procedure: hiHep Bioartificial Liver Support System — Continuous treatment with the hiHep bioartificial liver support system for a minimum of 3 days to a maximum of 14 days. The subject's ultrafiltrated blood is circulated through 4 cartridges. The parameter is set to Circuit 1：120-200ml/min；Circuit 2：30-50ml/min；Circuit 3：200 ml/min.
  Arms: Experimental group
Procedure: Standard care for ALF — A standard of care for subjects with acute liver failure.
  Arms: Control group

SUMMARY:
This study tend to evaluate safety and efficacy of hiHep bioartificial liver support system in treating acute liver failure.

DETAILED DESCRIPTION:
Liver damage remains a life-threatening syndrome. With the increasing number of patients awaiting transplantation, efforts have been made to develop extracorporeal methods to support or replace the function of the failing organ. A bioartificial liver support system has to provide the main functions of the liver: detoxification, synthesis, and regulation. It may prolonger the expected survival time of acute liver failure patients. Direct reprogramming of fibroblasts to hepatic lineages could offer a new type of solution to bioartificial liver support system. The investigators have already generated human induced hepatocytes (hiHeps) from fibroblasts by lentiviral expression of FOXA3, HNF1A, and HNF4A. hiHeps express hepatic gene programs, can be expanded in vitro, and display functions characteristic of mature hepatocytes, including cytochrome P450 enzyme activity and biliary drug clearance. hiHeps can restore the liver function and prolong survival. This study tends to evaluate safety and efficacy of hiHep bioartificial liver support system in treating acute liver failure.

ELIGIBILITY:
Inclusion Criteria:

* Weight more than 45 kg;
* Age more than 18;
* Diagnosis of ALF;
* Subjects must not be listed for transplant at the time of Enrollment or, if listed, in the opinion of the Investigator are unlikely to be transplanted within 72 hours;

Exclusion Criteria:

* Acute clinical symptoms that are likely to result in death within 48 hours;
* Presence of sepsis or septic shock;
* Concomitant disease including chronic congestive heart failure, severe vascular disease, emphysema, AIDS, cancer;
* Portal hypertension;
* Liver dysfunction due to trauma;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival of ALF subjects | Study Day 1 through Study Day 28
  Overall survival in subjects with acute liver failure will be summarized and compared with control subjects through Study Day 28.

SECONDARY OUTCOMES:
Complication rate | Study Day 1 through Study Day 60
  Proportion of subjects who suffer complications caused by bioartificial liver support system

CONTACTS AND LOCATIONS:
Overall Officials: Shaolin Ma, MD., Principal Investigator — Department of ICU, Shanghai East Hospital, School of Medicine, Tongji University

IPD SHARING:
Plan to Share IPD: No